CLINICAL TRIAL: NCT04573946
Title: VITamin D and OmegA-3 TriaL: Interrelationship of Vitamin D and Vitamin K on Bone
Brief Title: VITamin D and OmegA-3 TriaL: Interrelationship of Vitamin D and Vitamin K on Bone (VITAL)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Meryl LeBoff, Director of Skeletal Health and Osteoporosis Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012P000560-1; 2R01AR059775-06A1 (NIH); 5R01AR060574-03 (NIH)
Record Dates: First submitted 2020-09-01; First posted 2020-10-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Bone Density; Bone Health; Fractures
Keywords: Vitamin D; Vitamin K
MeSH Terms: conditions — Fractures, Bone | interventions — Fatty Acids, Omega-3; Fish Oils; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D placebo + fish oil placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3 placebo; Drug: Omega-3 fatty acids (fish oil)
- Vitamin D + fish oil placebo (Active Comparator)
  Interventions: Dietary Supplement: Fish oil placebo; Dietary Supplement: Vitamin D3
- Vitamin D + fish oil (Active Comparator)
  Interventions: Drug: Omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 placebo — Vitamin D placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo
Dietary Supplement: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo
Drug: Omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day.
  Other Names: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo

SUMMARY:
Vitamin D supplements are widely promoted for bone health. Both vitamin D and vitamin K are important for deposition of calcium in bone, but little is known about the relationship of vitamin K status and bone health.

DETAILED DESCRIPTION:
The goal of VITAL: Interrelationship of Vitamin D and Vitamin K on Bone is to test whether vitamin K status is associated with incident fractures in a case-cohort design or modifies the randomized effects of vitamin D supplementation vs. placebo on 2-year changes in bone density and structure outcomes.

ELIGIBILITY:
Inclusion:

- Participants in VITAL (NCT 01169259) study who met the following criteria of the parent trial are eligible to participate in this ancillary study:

* be men aged 50 years and older or women aged 55 years and older
* have no history of cardiovascular disease or cancer (excluding non-melanoma skin cancer)
* have none of the following: allergy to soy or fish, hypercalcemia, renal failure or dialysis, severe liver disease, hypo- or hyperparathyroidism, sarcoidosis or other granulomatous diseases, or any other serious illnesses
* consume ≤ 1200 mg/d of calcium for the duration of the trial
* consume ≤ 800 IU of vitamin D for duration of the trial
* refrain from taking fish oil supplements for the duration of the trial

Exclusion:

- For aims 2 and 3, those who are using bisphosphonates currently or within the past 2 years, or other bone-active medications currently or within the past year are not eligible for this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25871 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Fractures | 2 years
  The effect of low vitamin K status (with or without vitamin D supplementation) on the number of new total, non-vertebral and hip fractures.

SECONDARY OUTCOMES:
Change in Areal Bone Density | 2 years
  The effect of low vitamin K status (with or without vitamin D supplementation) on changes in areal bone density at the spine and hip between baseline and two years post-randomization.
Change in Volumetric Bone Mineral Density | 2 years
  The effect of low vitamin K status (with or without vitamin D supplementation) on changes in total, trabecular and cortical volumetric bone mineral density (vBMD) between baseline and two years post-randomization.
Change in Cortical Thickness | 2 years
  The effect of low vitamin K status (with or without vitamin D supplementation) on changes in cortical thickness assessed by peripheral quantitative computed tomography (pQCT) between baseline and two years post-randomization.
Change in Bone Strength | 2 years
  The effect of low vitamin K status (with or without vitamin D supplementation) on changes in bone strength measures assessed by peripheral quantitative computed tomography (pQCT) between baseline and two years post-randomization.
Change in Trabecular Bone Score | 2 years
  The effect of low vitamin K status (with or without vitamin D supplementation) on changes in trabecular bone score between baseline and two years post-randomization.
Concentration of Urine Calcium | 2 years
  The effect of low vitamin K status (with or without vitamin D supplementation) on change in urine calcium excretion between baseline and two years post-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Meryl S LeBoff, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] LeBoff MS, Yue AY, Copeland T, Cook NR, Buring JE, Manson JE. VITAL-Bone Health: rationale and design of two ancillary studies evaluating the effects of vitamin D and/or omega-3 fatty acid supplements on incident fractures and bone health outcomes in the VITamin D and OmegA-3 TriaL (VITAL). Contemp Clin Trials. 2015 Mar;41:259-68. doi: 10.1016/j.cct.2015.01.007. Epub 2015 Jan 24. PMID 25623291
- [Background] Donlon CM, LeBoff MS, Chou SH, Cook NR, Copeland T, Buring JE, Bubes V, Kotler G, Manson JE. Baseline characteristics of participants in the VITamin D and OmegA-3 TriaL (VITAL): Effects on Bone Structure and Architecture. Contemp Clin Trials. 2018 Apr;67:56-67. doi: 10.1016/j.cct.2018.02.003. Epub 2018 Feb 23. PMID 29408561
- [Background] Goldman AL, Donlon CM, Cook NR, Manson JE, Buring JE, Copeland T, Yu CY, LeBoff MS. VITamin D and OmegA-3 TriaL (VITAL) bone health ancillary study: clinical factors associated with trabecular bone score in women and men. Osteoporos Int. 2018 Nov;29(11):2505-2515. doi: 10.1007/s00198-018-4633-3. Epub 2018 Jul 18. PMID 30022253
- [Background] LeBoff MS, Chou SH, Murata EM, Donlon CM, Cook NR, Mora S, Lee IM, Kotler G, Bubes V, Buring JE, Manson JE. Effects of Supplemental Vitamin D on Bone Health Outcomes in Women and Men in the VITamin D and OmegA-3 TriaL (VITAL). J Bone Miner Res. 2020 May;35(5):883-893. doi: 10.1002/jbmr.3958. Epub 2020 Jan 30. PMID 31923341
- See also: VITAL Study Website — http://www.vitalstudy.org/